CLINICAL TRIAL: NCT01394562
Title: Multicentre, Prospective, Randomised, 2-arm Study to Assess the Impact of Ferric Carboxymaltose on Exercise Capacity in Chronic Heart Failure Patients With Iron Deficiency
Brief Title: Effect of Ferric Carboxymaltose on Exercise Capacity in Patients With Iron Deficiency and Chronic Heart Failure
Acronym: EFFECT-HF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vifor Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FER-CARS-04; 2011-000603-40 (EudraCT Number)
Record Dates: First submitted 2011-07-12; First posted 2011-07-14 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2015-12

CONDITIONS: Iron Deficiency; Chronic Heart Failure
MeSH Terms: conditions — Iron Deficiencies | interventions — ferric carboxymaltose; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ferinject (ferric carboxymaltose) (Experimental)
  Interventions: Drug: Ferinject (ferric carboxymaltose)
- Standard of Care (Other): Standard of care. IV iron is not permitted
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: Ferinject (ferric carboxymaltose) — Subjects will receive ferric carboxymaltose intravenously on Day 0, Week 6, and Week 12
  Arms: Ferinject (ferric carboxymaltose)
Other: Standard of Care — Subjects randomised to Standard of Care may receive oral iron at Investigator's discretion however patients will not be permitted to receive IV iron
  Arms: Standard of Care

SUMMARY:
The purpose of this study is to confirm that treatment with IV ferric carboxymaltose improves exercise capacity, physical functioning and quality of life in patients with iron deficiency and chronic heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Iron deficient subjects with stable chronic heart failure (CHF) (NYHA II-III) on optimal background therapy for CHF
* Reduced exercise capacity
* Reduced left ventricular ejection fraction
* At least 18 years of age and with written informed consent prior to any study specific procedures

Exclusion Criteria:

* Erythropoietin stimulating agent (ESA) use, IV iron therapy, and/or blood transfusion in previous 6 weeks prior to randomisation
* Exercise training program(s) in the 3 months prior to screening or planned in the next 6 months
* Chronic liver disease and/or elevated liver enzymes
* Vitamin B12 and/or serum folate deficiency
* Subject is not using adequate contraceptive precautions during the study
* No other significant cardiac or general disorder that would compromise participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2011-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in Peak VO2 (mL/kg/min) from baseline to Week 24 | Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Dirk van Veldhuisen, MD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Derived] van Veldhuisen DJ, Ponikowski P, van der Meer P, Metra M, Bohm M, Doletsky A, Voors AA, Macdougall IC, Anker SD, Roubert B, Zakin L, Cohen-Solal A; EFFECT-HF Investigators. Effect of Ferric Carboxymaltose on Exercise Capacity in Patients With Chronic Heart Failure and Iron Deficiency. Circulation. 2017 Oct 10;136(15):1374-1383. doi: 10.1161/CIRCULATIONAHA.117.027497. Epub 2017 Jul 12. PMID 28701470